CLINICAL TRIAL: NCT02272387
Title: Is Vitamin D Insufficiency and Deficiency Associated With Antepartum and Postpartum Depression?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment and limited research staffing
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-0223
Record Dates: First submitted 2014-10-16; First posted 2014-10-22 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Depression; Postpartum Depression
MeSH Terms: conditions — Depression; Depression, Postpartum | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 (cholecalciferol) treatment (Active Comparator): 50,000 IU vitamin D3 (cholecalciferol) tablet weekly x 8 weeks plus prenatal vitamin (400 IU vitamin D)
  Interventions: Dietary Supplement: Vitamin D3 (Cholecalciferol)
- Vitamin D placebo (Placebo Comparator): Placebo tablet (appearance same as active vitamin D) plus prenatal vitamin (400IU vitamin D)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (Cholecalciferol)
  Arms: Vitamin D3 (cholecalciferol) treatment
Other: Placebo
  Arms: Vitamin D placebo

SUMMARY:
Our primary aim is to evaluate whether Vitamin D deficiency causes depressive symptoms in antepartum and postpartum depression and whether early correction of Vitamin D deficiency improves these symptoms.

Our secondary aims evaluate maternal and fetal outcomes including antepartum, intrapartum, and immediate postpartum complications. We are also evaluating the effectiveness of a common vitamin D treatment regimen used outside of pregnancy.

DETAILED DESCRIPTION:
Our study recruitment will be at a single center in our pregnant private and clinic population. We will recruit eligible pregnant women 20 weeks 0 days or less. On study entry, patients will complete a demographic survey, vitamin D exposure survey, and an Edinburgh Postnatal Depression Score (EPDS) questionnaire. Baseline vitamin D levels will be obtained using a 25 OH D (vitamin D) assay.

Women found to be vitamin D deficient/insufficient will be approached for randomization to vitamin D3 (Cholecalciferol) 50,000 IU/week x 8 weeks + prenatal vitamin versus placebo + prenatal vitamin. A repeat 25 OH D sample plus a vitamin D exposure and EPDS questionnaires will be obtained between 24-28 weeks gestation upon completing treatment. All patients will then be kept on maintenance vitamin D until delivery (total vitamin D 800IU/day which includes prenatal vitamin). Delivery 25 OH D samples will be collected on all women. At delivery, these women will also complete vitamin D exposure and EPDS questionnaires. Maternal and fetal outcome data will be collected on all patients.

As for vitamin D sufficient patients, they will be followed with vitamin D exposure and EPDS questionnaires at 24-28 weeks and delivery. A 25 OH D sample will be obtained at delivery for these women. Maternal and fetal outcome data will be obtained.

For vitamin D deficient women declining randomization, they will be given vitamin D repletion based on their preference after counseling. We will continue to follow their questionnaires and outcomes similarly to the vitamin D sufficient group.

ELIGIBILITY:
Inclusion Criteria:

* Evaluation at Roosevelt Hospital (Receiving prenatal care with St Luke's Roosevelt Hospital center private physicians and clinic) by 20w0d gestation.
* Planned delivery at Roosevelt Hospital Labor & Delivery
* English or Spanish speaking

Exclusion Criteria:

* Non-english or non-spanish speaking
* Currently on anti-depressants/mood stabilizing medications
* Medical comorbidities affecting vitamin D absorption or metabolism:Bone disease (osteoporosis, osteomalacia); Malabsorption disorders (cystic fibrosis, inflammatory bowel disease, roux-en-y bariatric surgery); Chronic kidney disease; Severe liver disease; Granuloma forming disorders (active tuberculosis, sarcoidosis);Parathyroid disease; Lymphoma; HIV on HAART medication; anti-seizure medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-04-14 (Actual); Study Completion 2016-04-14 (Actual)

PRIMARY OUTCOMES:
Antepartum and Postpartum Depressive symptoms | 9 months
  We will be using an Edinburgh Postnatal Depression Scale (EPDS) questionnaire to monitor depressive symptoms.

SECONDARY OUTCOMES:
Maternal morbidities | Antepartum and Delivery
  Composite maternal complications: preeclampsia, GDM, delivery complications, chorioamnionitis, etc.
Fetal morbidities | Antepartum and delivery
  Composite outcomes: SGA, IUGR, low apgars, low cord gases, hydramnios, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Roosevelt Hospital, New York, New York, United States